CLINICAL TRIAL: NCT00271141
Title: Multifunctional Substrate for Early Detection of Oxidative Stress Susceptibility and Application to Parkinson's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Collaborators: Technion, Israel Institute of Technology (Other)
Other Study IDs: hy11/2005
Record Dates: First submitted 2005-12-29; First posted 2005-12-30 (Estimated); Last update posted 2005-12-30 (Estimated); Status verified 2005-12

CONDITIONS: Parkinson's Disease; Oxidative Stress
Keywords: Parkinson's disease; Oxidative stress; Marker
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
The proposed work is based on the detection of a novel molecule for sensitivity to oxidative stress in humans in venous blood

DETAILED DESCRIPTION:
Since alterations in mitochondrial functions in platelets and lymphocytes have been detected in Parkinson's disease we plan to monitor the metabolism a a new molecule (LTG) in the blood samples of Parkinson's disease patients and compare them to controls. We shall use 10 cc of venous blood and analyze serum, white blood cells and platelets. We shall not extract nor use DNA.The main purpose is to develop a marker for Parkinson's disease in venous blood.

ELIGIBILITY:
Inclusion Criteria:

Parkinson's disease Healthy control -

Exclusion Criteria:

None -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2005-05; Study Completion 2015-12

CONTACTS AND LOCATIONS:
Overall Officials: Rivka Inzelberg, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel